CLINICAL TRIAL: NCT02910063
Title: A Phase 2/3 Multi-center Study to Evaluate the Safety and Efficacy of Blinatumomab in Subjects With Relapsed/Refractory Aggressive B-Cell Non Hodgkin Lymphoma
Brief Title: Study to Evaluate Safety and Efficacy of Blinatumomab in Subjects With Relapsed/Refractory (R/R) Aggressive B-Cell NHL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20150292; 2016-002044-16 (EudraCT Number)
Record Dates: First submitted 2016-08-30; First posted 2016-09-21 (Estimated); Results first posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: B-Cell Non Hodgkin Lymphoma
Keywords: Relapsed/Refractory Aggressive B-Cell Non Hodgkin Lymphoma; Blinatumomab; Leukemia; Standard of Care; SOC; Cancer; Chemotherapy
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence; Leukemia; Neoplasms | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blinatumomab (Experimental): Blinatumomab is administered as a continuous intravenous infusion (CIVI). A single cycle of blinatumomab is continuous infusion with step dosing of 9 µg/day x 7 days, 28 µg/day x 7 days, and 112 µg/days until the end of the cycle.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab monotherapy
  Other Names: AMG 103; Blincyto

SUMMARY:
This is a phase 2/3 open label, multicenter trial testing blinatumomab monotherapy for the treatment of subjects with Relapsed/Refractory (R/R) aggressive B-NHL not achieving CMR after 2 cycles of standard platinum-based chemotherapy regimens administered as S1. This study incorporates multiple interim analyses for futility, efficacy, and unblinded sample-size re-estimation. In the phase 3 part of the study, blinatumomab will be compared to Investigator's Choice chemotherapy.

In March 2019, decision made to not proceed with phase 3.

DETAILED DESCRIPTION:
This is a phase 2/3 open label, multicenter trial testing blinatumomab monotherapy for the treatment of subjects with R/R aggressive B-NHL not achieving CMR after standard platinum-based chemotherapy regimens administered as S1. This study incorporates multiple interim analyses for futility, efficacy, and unblinded sample-size re-estimation. In the phase 3 part of the study, blinatumomab will be compared to IC chemotherapy.The phase 2 component of the study will consist of up to a 28-day screening period, approximately 70 to 112 days of study treatment, a 30-day (+/- 3days) safety follow up, and long-term follow up that will conclude with the final analysis of the phase 3 component, estimated at 30 months after initiation of the phase 3 component. For the phase 3 component, the study will consist of up to a 28-day screening period, a treatment period of up to approximately 168 days, a 30-day safety follow-up visit, and long-term follow up. Long-term follow up will conclude with the final analysis.In the phase 2 component, enrolled subjects will receive blinatumomab monotherapy. In the phase 3 component, enrolled subjects will be randomized in a 1:1 ratio to blinatumomab or IC chemotherapy.

In March 2019, decision made to not proceed with phase 3.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven aggressive B-cell Non-Hodgkin Lymphoma (B-NHL), including diffuse large B-cell lymphoma (DLBCL) not otherwise specified (NOS), follicular lymphoma Grade 3B, PMBCL, T-cell rich B-cell lymphoma, or DLBCL that represents transformation of indolent non-Hodgkin's Lymphoma (NHL), (including follicular, marginal zone, and lymphoplasmacytoid lymphoma) excluding chronic lymphocytic leukemia or Hodgkin Lymphoma. The following histologies are not eligible:

  * Lymphoblastic lymphoma
  * Burkitt lymphoma
  * Mantle cell lymphoma Any histologies not specifically mentioned must be discussed with medical monitor.
* Refractory (no prior CR/CMR) or relapsed (prior CMR) following front line treatment of standard multiagent chemotherapy containing an anthracycline AND an approved anti-CD20 agent. For subjects with refractory disease and who have received radiotherapy, PET positivity should be demonstrated no less than 6 weeks after the last dose of radiotherapy
* Biopsy proven confirmation of relapsed disease.
* Received a minimum of 2 cycles of standard of care platinum-based chemotherapy in the S1 setting and had a response of progressive metabolic disease (PMD), no metabolic response (NMR), partial metabolic response (PMR) as centrally assessed by PET-/ CT scan or received at least 1 cycle of S1 chemotherapy and had evidence of PMD as centrally assessed. A pre-salvage scan is required to be submitted to the central reader if a subject had only 1 cycle of pre-salvage chemotherapy.
* Radiographically measurable disease with a demarcated nodal lesion at least 1.5 cm in its largest dimension or a target extranodal lesion at least 1.0 cm in its largest dimension
* Eastern Cooperative Oncology Group performance status less than or equal to 2
* Intention to proceed to high dose chemotherapy (HDT) and autologous hematopoietic stem cell transplant (HSCT)
* Laboratory parameters:

Hematology:

* Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L
* Platelets ≥ 75 x 10^9/L

Chemistry:

* Creatinine clearance ≥ 50 mL/min
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 3X upper limit of normal (ULN)
* Total bilirubin (TBL) < 2x ULN (unless Gilbert's disease or if liver involvement with lymphoma)

Exclusion Criteria:

* CMR following S1 chemotherapy
* Treatment within 30 days prior to randomization with another investigational device or drug study (ies).
* Prior anti-CD19-directed therapies
* Prior HDT with autologous HSCT
* Prior allogeneic HSCT
* Clinically relevant central nervous system (CNS) pathology such as epilepsy, paresis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
* Evidence of CNS involvement by NHL
* Known infection with human immunodeficiency virus or chronic infection with hepatitis B virus (hepatitis B surface antigen positive) or hepatitis C virus (anti hepatitis C virus positive)
* History of malignancy other than B-NHL within the past 3 years with the exception of:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment
  * Adequately treated non-melanoma skin cancer or lentigo maligna
  * Adequately treated cervical carcinoma in situ
  * Adequately treated breast ductal carcinoma in situ
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer
  * Adequately treated urothelial papillary non-invasive carcinoma or carcinoma in situ
* Known sensitivity to immunoglobulins or any of the components to be administered during dosing.
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required procedures.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Female subjects who are pregnant or breastfeeding or planning to become pregnant or breastfeed, or of childbearing potential unwilling to use an effective method of contraception while receiving, and for an additional 48 hours after the last dose of blinatumomab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (30):
- United States (4):
  - Research Site, Duarte, California
  - Research Site, Baltimore, Maryland
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Greenville, South Carolina
- Australia (5):
  - Research Site, St Leonards, New South Wales
  - Research Site, Herston, Queensland
  - Research Site, Melbourne, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Murdoch, Western Australia
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
- Research Site, Montreal, Quebec, Canada
- Italy (7):
  - Research Site, Bergamo
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Udine
- Research Site, San Juan, Puerto Rico
- Spain (6):
  - Research Site, Córdoba, Andalusia
  - Research Site, Valladolid, Castille and León
  - Research Site, Barcelona, Catalonia
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Madrid
  - Research Site, Murcia
- United Kingdom (3):
  - Research Site, Bristol
  - Research Site, Nottingham
  - Research Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Coyle L, Morley NJ, Rambaldi A, Mason KD, Verhoef G, Furness CL, Zhang A, Jung AS, Cohan D, Franklin JL. Open-Label, phase 2 study of blinatumomab as second salvage therapy in adults with relapsed/refractory aggressive B-cell non-Hodgkin lymphoma. Leuk Lymphoma. 2020 Sep;61(9):2103-2112. doi: 10.1080/10428194.2020.1759055. Epub 2020 Jun 16. PMID 32546071
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 19 research centers in Australia, Belgium, Italy, Spain, the United Kingdom, and the United States from 23 January 2017 to 15 January 2018.
Pre-assignment Details: Phase 3 part of the study was not initiated after Phase 2 data was reviewed. No participants were screened or enrolled for Phase 3.
Groups:
- Phase 2: Blinatumomab: Participants entered a single 70-day dose step cycle, and received a total of 56 days of blinatumomab continuous infusion which was administered as 7 days at 9 microgram (μg)/day, 7 days at 28 μg/day, and 42 days at 112 μg/day, followed by a treatment-free period of 14 days.
  Eligible participants could then enter an optional Cycle 2, 2 to 4 weeks after the end of the previous cycle. The optional Cycle 2 consisted of a 28-day cycle of blinatumomab continuous infusion administered as 7 days at 9 μg/day, 7 days at 28 μg/day, and 14 days at 112 μg/day.
- Phase 3: Blinatumomab: Participants were to enter a single 70-day dose step cycle, and received a total of 56 days of blinatumomab continuous infusion which was administered as 7 days at 9 microgram (μg)/day, 7 days at 28 μg/day, and 42 days at 112 μg/day, followed by a treatment-free period of 14 days.
  In March 2019, the decision made to not proceed with Phase 3 and no participants were enrolled. No data is available for Phase 3.
- Phase 3: Investigator's Choice (IC) Chemotherapy: Participants were to receive standard of care (SOC) chemotherapy per investigator´s choice.
  In March 2019, the decision was made to not proceed with Phase 3 and no participants were enrolled. No data is available for Phase 3.
Period: Phase 2
Arm/Group | Phase 2: Blinatumomab | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Started | 41 | 0 (Participants in this Phase 3 arm were not included in the Phase 2 period.) | 0 (Participants in this Phase 3 arm were not included in the Phase 2 period.)
Started Cycle 1 | 41 | 0 | 0
Started Optional Cycle 2 | 4 | 0 | 0
Completed | 13 | 0 | 0
Not Completed | 28 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Death | 24 | 0 | 0
Period: Phase 3
Arm/Group | Phase 2: Blinatumomab | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Started | 0 (Participants in this Phase 2 arm were not included in the Phase 3 period.) | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All participants who received blinatumomab.
Arm/Group | Phase 2: Blinatumomab
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 38
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 2: Percentage of Participants Who Achieved Complete Metabolic Response (CMR)
Description: Complete metabolic response (CMR) was determined by central radiographic assessment of positron emission tomography and computed tomography (PET/CT) scans using the Lugano Classification.
Time Frame: Up to 12 weeks after first dose of blinatumomab
Population: FAS: All participants who received blinatumomab.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Blinatumomab
Number analyzed (Participants) | 41
Percentage of participants | 22.0 [10.6 to 37.6]

2. Primary Outcome: Phase 3: Number of Participants Who Achieved Complete Metabolic Response (CMR)
Description: as for outcome 1
Time Frame: Up to 12 weeks after first dose of study treatment
Population: No data is available for Phase 3. In March 2019, the decision was made to not proceed with Phase 3 and no participants were enrolled.
Arm/Group | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until death due to any cause.
  OS was calculated using Kaplan-Meier estimates.
Time Frame: From randomization until the end of study, up to 30 months
Population: No data is available for Phase 3. In March 2019, the decision made to not proceed with Phase 3 and no participants were enrolled.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Blinatumomab
Number analyzed (Participants) | 41
Months | 11.2 [5.9 to NA] — Upper limit was not reached.

4. Secondary Outcome: Phase 2: Objective Response Rate (ORR)
Description: ORR is inclusive of all participants who achieved CMR or those who achieved partial metabolic response (PMR), as determined by central radiographic assessment of PET/CT scans using the Lugano Classification.
Time Frame: Up to 12 weeks after first dose of blinatumomab
Population: FAS: All participants who received blinatumomab.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Blinatumomab
Number analyzed (Participants) | 41
Percentage of participants | 36.6 [22.1 to 53.1]

5. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS was defined as the time from start of treatment with blinatumomab until the date of diagnosis of progression of lymphoma, or date of death, whichever is earliest. PFS was estimated using Kaplan-Meier method.
Time Frame: From first dose of blinatumomab until the end of study, up to 30 months
Population: FAS: All participants who received blinatumomab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Blinatumomab
Number analyzed (Participants) | 41
Months | 2.9 [2.3 to 5.3]

6. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR was calculated only for participants who achieve a response (CMR or PMR). The duration was calculated from the date a response, CMR or PMR, was first achieved until the earliest date of a disease assessment indicating disease progression or death, whichever occured first. DOR was estimated using Kaplan-Meier method.
Time Frame: From first dose of blinatumomab up to 12 weeks
Population: Full Analysis Set (FAS): All participants who received blinatumomab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Blinatumomab
Number analyzed (Participants) | 41
Months | 6.1 [2.5 to 10.7]

7. Secondary Outcome: Phase 2: Percentage of Participants Who Experienced Successful Mobilization
Description: Successful mobilization rate was defined as the percentage of participants who initiated mobilization while in remission and without any other anti-tumor therapy where the mobilization procedure had an outcome of 'Successful'. Successful mobilization was dictated by institutional standards and defined when the target cell dose was no less than 2 x 10^6 CD34+ cells/kg.
Time Frame: From first dose of blinatumomab until the end of study, up to 30 months
Population: Responder Analysis Set: All participants who had a CMR or PMR per central review during the first 12 weeks after initiation of blinatumomab.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Blinatumomab
Number analyzed (Participants) | 15
Percentage of participants | 40.0 [16.3 to 67.7]

8. Secondary Outcome: Phase 2: Percentage of Participants Who Had Allogeneic or Autologous Post-baseline Hematopoietic Stem Cell Transplant (HSCT)
Description: The percentage of responders per investigator's review (participants who achieved either CMR or PMR during the treatment) who have undergone allogeneic (allo) HSCT or autologous (auto) HSCT while in remission and without any other anti-cancer treatment.
Time Frame: From baseline HSCT until the end of study, up to 30 months
Population: FAS: All participants who received blinatumomab.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Blinatumomab
Number analyzed (Participants) | 41
Percentage of participants
  AlloHSCT | 6.7 [0.2 to 31.9]
  AutoHSCT | 53.3 [26.6 to 78.7]

9. Secondary Outcome: Phase 2: Cumulative Incidence Function Estimate of 100-day Mortality After HSCT Presented as Percentage of Participants That Died Not Due to Relapse, With Relapse and Death Due to Relapse as Competing Events
Description: Non-relapse mortality rate at 100 days after HSCT was calculated as the percentage of participants who died not due to relapse. Only participants who achieved a response per investigator's review and underwent autoHSCT are included.
Time Frame: 100 days after HSCT
Population: AutoHSCT Analysis Set: All participants who achieved a response and underwent autoHSCT while in remission and without any other anti-cancer treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Blinatumomab
Number analyzed (Participants) | 9
Percentage of participants | 0.0 [0.0 to 0.0]

10. Secondary Outcome: Phase 2: Blinatumomab Steady State Concentrations (Css)
Description: Pharmacokinetic (PK) parameters were estimated by non compartmental analysis. The Css of blinatumomab was summarized as the observed concentrations collected after at least 24 hours after the start of continuous IV infusion or start of dose step, where appropriate.
Time Frame: Pre-dose on Day 1, and post-dose on Days 2, 9 and 16 of Cycle 1 (Cycle 1 was 70 days)
Population: PK analysis Set: All subjects who received blinatumomab at each individual dose and had at least one PK sample collected.
Measure: Mean (Standard Deviation); unit: Picograms/millilter (pg/mL)
Groups:
- Phase 2: Blinatumomab 9 µg/Day: All participants who received blinatumomab 9 µg/day continuous infusion which was administered for 7 days of in Week 1 of Cycle 1 (Cycle 1 was 70 days in length).
- Phase 2: Blinatumomab 28 µg/Day: All participants who received blinatumomab 28 µg/day continuous infusion which was administered for 7 days in Week 2 of Cycle 1 (Cycle 1 was 70 days in length).
- Phase 2: Blinatumomab 112 µg/Day: All participants who received blinatumomab 112 µg/day continuous infusion which was administered for 7 days in Week 3 of Cycle 1 (Cycle 1 was 70 days in length).
Arm/Group | Phase 2: Blinatumomab 9 µg/Day | Phase 2: Blinatumomab 28 µg/Day | Phase 2: Blinatumomab 112 µg/Day
Number analyzed (Participants) | 41 | 38 | 32
Picograms/millilter (pg/mL) | 249 (200) | 804 (513) | 3470 (3700)

11. Secondary Outcome: Phase 2: Blinatumomab Clearance (CL)
Description: Serum blinatumomab CL was calculated as CL=R0/Css,DN; where R0 is the infusion rate (μg/hr) and Css,DN is the dose normalized average Css. For the CL calculation, the Css,DN was normalized to the 112 μg/day dose in which the value of dose in units of μg/hr was used for the infusion rate.
Time Frame: Pre-dose on Day 1, and post-dose on Days 2, 9 and 16 of Cycle 1 (Cycle 1 was 70 days)
Population: PK analysis Set: All subjects who received any infusion of blinatumomab and had at least one PK sample collected.
Measure: Mean (Standard Deviation); unit: Liter/hour (L/hr)
Arm/Group | Phase 2: Blinatumomab
Number analyzed (Participants) | 41
Liter/hour (L/hr) | 1.78 (0.747)

12. Secondary Outcome: Phase 2: Half-life of Blinatumomab
Time Frame: Pre-dose on Day 1, and Days 2, 9 and 16 of Cycle 1 (Cycle 1 was 70 days)
Population: Blinatumomab half-life was not reported as the serum blinatumomab concentration data collected for PK assessments did not support its estimation. This is in adherence with the considerations for reporting of PK assessments as detailed in Protocol Section 10.6.
Arm/Group | Phase 2: Blinatumomab
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase 2: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: Treatment-emergent adverse events were events with an onset after the administration of the first dose of blinatumomab.
  TEAEs were graded using the Common Terminology Criteria for Adverse Events (CTCAE).
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limited age appropriate instrumental activities of daily life (ADL).
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolonged hospitalization indicated; disabling; limited self care ADL.
  Grade 4 Life-threatening consequences; urgent interventions indicated.
Time Frame: From first dose of blinatumomab until 30 days after last dose. The maximum treatment duration for blinatumomab was 114 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Blinatumomab
Number analyzed (Participants) | 41
Participants
  TEAEs | 41
  Grade ≥ 2 TEAEs | 37
  Grade ≥ 3 TEAEs | 29
  Grade ≥ 4 TEAEs | 12
  Serious TEAEs | 20
  TEAEs leading to discontinuation of blinatumomab | 7
  TEAEs leading to interruption of blinatumomab | 13
  Fatal TEAEs | 7

14. Secondary Outcome: Phase 3: Objective Response Rate (ORR)
Time Frame: Up to 12 weeks after first dose of study treatment
Population: as for outcome 3
Arm/Group | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Phase 3: Progression Free Survival (PFS)
Time Frame: From first dose of study treatment until the end of study, up to 30 months
Population: as for outcome 3
Arm/Group | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Phase 3: Duration of Response (DOR)
Time Frame: From first dose of study treatment up to 12 weeks
Population: as for outcome 3
Arm/Group | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Phase 3: Percentage of Participants Who Experienced Successful Mobilization
Time Frame: From baseline until the end of study, up to 30 months
Population: as for outcome 3
Arm/Group | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Phase 3: Percentage of Participants Who Had Allogeneic or Autologous Post-baseline Hematopoietic Stem Cell Transplant (HSCT)
Time Frame: From baseline HSCT until the end of study, up to 30 months
Population: as for outcome 3
Arm/Group | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Phase 3: Percentage of Participants Who Died Within 100 Days After Hematopoietic Stem Cell Transplantation (HSCT) That Was Not Due to Relapse
Time Frame: 100 days after HSCT
Population: as for outcome 3
Arm/Group | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Phase 3: Change From Baseline in Patient Reported Clinical Outcome Assessments Quality of Life (QOLCOA) Scores
Time Frame: Up to 30 days after last dose after study treatment
Population: as for outcome 3
Arm/Group | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Phase 3: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Time Frame: From first dose of study treatment until 30 days after last dose
Population: as for outcome 3
Arm/Group | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Phase 3: Serum Blinatumomab Steady State Concentration (Css)
Time Frame: 24 hours after first dose of blinatumomab
Population: as for outcome 3
Arm/Group | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Phase 3: Blinatumomab Clearance (CL)
Time Frame: Pre-dose on Day 1, and Days 2, 9 and 16 of Cycle 1 (Cycle 1 was 70 days)
Population: as for outcome 3
Arm/Group | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Phase 3: Half-life of Blinatumomab
Time Frame: Pre-dose on Day 1, and Days 2, 9 and 16 of Cycle 1 (Cycle 1 was 70 days)
Population: as for outcome 3
Arm/Group | Phase 3: Blinatumomab | Phase 3: Investigator's Choice (IC) Chemotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of blinatumomab until 30 days after last dose. The maximum treatment duration for blinatumomab was 114 days
Description: All-cause mortality, serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
  No data is available for Phase 3. In March 2019, decision made to not proceed with Phase 3 and no participants were enrolled. The data below is only inclusive of participants in Phase 2.
Arm/Group | Phase 2: Blinatumomab
All-Cause Mortality (participants affected / at risk) | 25/41
Serious Adverse Events (participants affected / at risk) | 20/41
Other Adverse Events (participants affected / at risk) | 29/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2: Blinatumomab (N=41)
Atrial fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Staphylococcal bacteraemia (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemiparesis (Nervous system disorders) | 1
Neurotoxicity (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2: Blinatumomab (N=41)
Anaemia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 3
Fatigue (General disorders) | 4
Oedema peripheral (General disorders) | 8
Pyrexia (General disorders) | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Aphasia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 10
Paraesthesia (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 9
Confusional state (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Hypotension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
Phase 3 part of the study was not initiated after Phase 2 data was reviewed. No participants were screened or enrolled for Phase 3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT02910063/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT02910063/SAP_001.pdf